CLINICAL TRIAL: NCT04526262
Title: Single-center, Open, Prospective, Single-arm, Feasibility, Investigator-initiated Trail for Assessment of Initial Efficacy and Safety of High Intensity Focused Ultrasound 'ExAblate 4000 Type 2' for Blood Brain Barrier Disruption in Patients With Alzheimer's Disease
Brief Title: Assessment of Initial Efficacy and Safety of High Intensity Focused Ultrasound 'ExAblate 4000 Type 2' for Blood Brain Barrier Disruption in Patients With Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2019-0095
Record Dates: First submitted 2020-08-19; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BBB disruption (Experimental): All participant in this arm will undergo 2 sessions of transcranial magnetic resonance guided focused ultrasound blood brain barrier disruption every 3 months.
  Interventions: Device: transcranial magnetic resonance guided focused ultrasound BBB disruption

INTERVENTIONS:
Device: transcranial magnetic resonance guided focused ultrasound BBB disruption — The ExAblate BBB disruption procedure will be performed with ExAblate 4000 type 2.0 system, and this will be performed twice every 3 months.

SUMMARY:
The proposed study is to evaluate initial efficacy and safety of the BBB disruption with transcranial MRI-guided focused ultrasound (ExAblate 4000 type 2.0) in patients with Alzheimer's disease.

This study iw designed as a prospective, single-site, single-aarm, nonrandomized study. Assessments will be made before and three months after 2 sessions of BBB disruption with radiologic, nuclear medicine imaging and neurophysiological examinations. Relative safety will be evaluated using a common description of Significant Clinical Complications for patients treated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 85 years, inclusive.
* Total score of 23 or less on the Korean version of Mini Mental state Exam (K-MMSE)
* FBB (18F-Florbetaben)-PET test result positive
* FDB (18F-Fluorodeoxyglucose)-PET test results suspected of Alzheimer disease-induced neurodegeneration
* Mild cognitive impairment or dementia caused by Alzheimer's disease
* A participant who has been given a drug at a stable dose for at least three months to improve symptoms of Alzheimer's disease
* Able to communicate during the ExAblate BBB disruption procedure
* Able and willing to give informed consent
* Able to attend all study visits

Exclusion Criteria:

* CGA-NPI (Caregiver-Administrated Neuropsychiatry Inventory) severity score of more than 2 points for any of "Delusion", "Hallucination" or "Agitation/Aggression"
* Known sensitivity/allergy or contraindications to MRI contrast agent(Gadovist®) or the ultrasound contrast agent (Definity®)
* Contraindications to MRI such as non-MRI compatible implanted devices.
* Any of the following items in MRI

  1. severe ischemic changes
  2. active or chronic infection/inflammation
  3. acute or chronic hemorrhage
  4. tumor/space occupying lesion
  5. meningeal enhancement
  6. intracranial hypotension
* More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
* Active seizure disorder or epilepsy (seizures despite medical treatment)
* History of a bleeding disorder, coagulopathy
* Cardiac disease or unstable hemodynamics
* Severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2
* Severe brain atrophy
* HIV (Human immunodeficiency virus) positive, who have a high probability of developing HIV encephalitis due to the influx of HIV in to the brain parenchyma
* Subjects with evidence of cranial or systemic infection
* A homozygosity of Apolipoprotein E allele (ApoE4) known to have a thin blood-brain barrier
* Positive pregnancy test (women of childbearing potential)
* A participant in other clinical trials or have experience in other clinical trials within 90 days from the screening date

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events safety profile | 6 months
  The type and severity of post-procedure adverse events will be assessed for overall safety. Safety of the BBBD procedure will be evaluated through patient examination and MRI assessements during the treatment and by their standard care of follow-up MRI scans and clinical visits.

SECONDARY OUTCOMES:
Efficacy of BBB disruption : evaluated by radiologic imaging | 6 months
  The efficacy of BBB disruption in Alzheimer's disease will be evaluated by radiologic, nuclear medicine imaging and neurophysiological examination.
Efficacy of BBB disruption : evaluated by nuclear medicine imaging | 6 months
  The efficacy of BBB disruption in Alzheimer's disease will be evaluated by radiologic, nuclear medicine imaging and neurophysiological examination.
Efficacy of BBB disruption : evaluated by neurophysiological examination | 6 months
  The efficacy of BBB disruption in Alzheimer's disease will be evaluated by radiologic, nuclear medicine imaging and neurophysiological examination.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Woo Chang, Principal Investigator — Severance Hospital
Locations (1):
- Department of Neurosurgery, Yonsei University College of Medici, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided